CLINICAL TRIAL: NCT04468464
Title: Quantitative Evaluation of Osteopathic Treatment in Temporomandibular Joint Disorders Using Magnetic Resonance Imaging
Acronym: TMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACorekci
Record Dates: First submitted 2020-07-06; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Temporomandibular Disorders, Articular Disc Disorder (Reducing or Non-Reducing); Osteopathy in Temporomandibular Disorders
Keywords: temporomandibular disorders, anterior disc displacement with reduction, MRI analyses, Osteopathy
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: Both groups receive splint treatment, but study group also receives osteopathic manual treatment
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Radiologist who evaluates the MRI results was blinded about the group of participants and also blinded about the diagnosis of the dentist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Occlusal Splint
  Interventions: Other: Occlusal Splint Treatment
- Study Group (Experimental): Osteopathic Manuel Therapy
  Interventions: Other: Occlusal Splint Treatment; Other: Osteopathic Manual Treatment

INTERVENTIONS:
Other: Occlusal Splint Treatment — Occlusal splint is used by a dentist during sleep or day time to protect the teeth and temporomandibular joint. Manufactured individually by the technicians according to the dentists measurement procedure.
Other: Osteopathic Manual Treatment — Osteopathy treats the body as a whole and applied by hands over the related structures of the body. TMJ, Cervical, Thoracal, Lumbar vertebra mobilization was applied as well as the fascial and visceral mobilization. Patients also used occlusal splint for 6 weeks during the intervention.
  Arms: Study Group

SUMMARY:
The aim of this study is to assess the impact of osteopathic manual treatment in patients with an anterior disc displacement over sleep and health quality, pain scores and the movement of the condyle and disc of the temporomandibular joint (TMJ) quantitatively.

DETAILED DESCRIPTION:
Patients with TMD will involve to this study. After having the diagnose in Yeditepe U. Dental Hospital patients will be sent to the Radiology Department. MRI images will be gathered in sagittal, coronal and axial plane for each patient before and after treatment. Volunteers will be divided into two groups; (1) splint therapy for 6 weeks, (2) splint therapy + osteopathy 2 times a week for 6 weeks randomly. At the end of the treatment, patients will be sent to Radiology for the second images. Health Survey and pain scores, Disc condyle angle, disc and condyle displacements will be measured and compared inter and intra groups.

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of TMD (anterior disc displacement)

Exclusion Criteria:

* Active orthodontic treatment
* Systemic diseases
* Oral or dental pathologies
* Dental implant placement
* Exodontia within 6 months
* Cranial and cervical trauma or surgery
* Taking antidepressant medication
* Contraindication of MRI scans

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Temporomandibular Joint Pain | 6 weeks after the first measurement
  10 point scale 0- no pain 10- severe pain
Change in TMJ MR images | 6 weeks after the first measurement
  Disc-condyle angle, disc and condyle positions were measured over TMJ images
Change in Mandibular Movements | 6 weeks after the first measurement
  Depression, Left and Right lateralization of the mandibula was measured by the caliper
Change in Cervical Movement | 6 weeks after the first measurement
  Cervical Region range of motions was measured by a goniometer

SECONDARY OUTCOMES:
Changes in bodily pain | 6 weeks after the first measurement
  10 point scale 0- no pain 10- severe pain

OTHER OUTCOMES:
Change in Life Quality score | 6 weeks after the first measurement
  A high score corresponds to a good quality of life
Change in sleep quality score | 6 weeks after the first measurement
  A high score corresponds to a low quality of the sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalamir, A., Pollard, H., Vitiello, A. L., & Bonello, R. (2007). Manual therapy for temporomandibular disorders: A review of the literature. Journal of Bodywork and Movement Therapies, 11(1), 84-90. https://doi.org/10.1016/j.jbmt.2006.07.003
- [Background] Kurita H, Kurashina K, Ohtsuka A, Kotani A. Change of position of the temporomandibular joint disk with insertion of a disk-repositioning appliance. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Feb;85(2):142-5. doi: 10.1016/s1079-2104(98)90416-4. PMID 9503446
- [Background] Gesslbauer C, Vavti N, Keilani M, Mickel M, Crevenna R. Effectiveness of osteopathic manipulative treatment versus osteopathy in the cranial field in temporomandibular disorders - a pilot study. Disabil Rehabil. 2018 Mar;40(6):631-636. doi: 10.1080/09638288.2016.1269368. Epub 2016 Dec 28. PMID 28029069